CLINICAL TRIAL: NCT01362374
Title: A Phase Ib, Open-label, Dose-escalation Study of the Safety and Pharmacology of Ipatasertib (GDC-0068) in Combination With Docetaxel, Fluoropyrimidine Plus Oxaliplatin, Paclitaxel, or Enzalutamide in Patients With Advanced Solid Tumors
Brief Title: Safety and Clinical Pharmacology of GDC-0068 in Combination With Docetaxel, Fluoropyrimidine Plus Oxaliplatin, Paclitaxel, or Enzalutamide in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAM4983g; GO27845 (Other: Hoffmann-La Roche); 2011-000782-13 (EudraCT Number)
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Fluorouracil; Docetaxel; enzalutamide; ipatasertib; Leucovorin; Oxaliplatin; Paclitaxel

ARMS (13):
- Arm A (Doc + Ipat 100mg) (Experimental): Participants received ipatasertib at a dose of 100 milligrams (mg) once daily for 14 consecutive days (beginning on Day 2) in combination with docetaxel on Day 1, in 21-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: Docetaxel; Drug: Ipatasertib
- Arm A (Doc + Ipat 200mg) (Experimental): Participants received ipatasertib at a dose of 200mg once daily for 14 consecutive days (beginning on Day 2) in combination with docetaxel on Day 1, in 21-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: Docetaxel; Drug: Ipatasertib
- Arm A (Doc + Ipat 400mg) (Experimental): Participants received ipatasertib at a dose of 400mg once daily for 14 consecutive days (beginning on Day 2) in combination with docetaxel on Day 1, in 21-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: Docetaxel; Drug: Ipatasertib
- Arm A (Doc + Ipat 600mg) (Experimental): Participants received ipatasertib at a dose of 600mg once daily for 14 consecutive days (beginning on Day 2) in combination with docetaxel on Day 1, in 21-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: Docetaxel; Drug: Ipatasertib
- Arm B (mFOLFOX + Ipat 100mg) (Experimental): Participants received ipatasertib at a dose of 100mg once daily for 7 consecutive days (beginning on Day 1) in combination with mFOLFOX6 chemotherapy (comprising of oxaliplatin, leucovorin, and 5-FU) on Day 1, in 14-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: 5-FU; Drug: Ipatasertib; Drug: Leucovorin; Drug: Oxaliplatin
- Arm B (mFOLFOX + Ipat 200mg) (Experimental): Participants received ipatasertib at a dose of 200mg once daily for 7 consecutive days (beginning on Day 1) in combination with mFOLFOX6 chemotherapy (comprising of oxaliplatin, leucovorin, and 5-FU) on Day 1, in 14-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: 5-FU; Drug: Ipatasertib; Drug: Leucovorin; Drug: Oxaliplatin
- Arm B (mFOLFOX + Ipat 400mg) (Experimental): Participants received ipatasertib at a dose of 400mg once daily for 7 consecutive days (beginning on Day 1) in combination with mFOLFOX6 chemotherapy (comprising of oxaliplatin, leucovorin, and 5-FU) on Day 1, in 14-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: 5-FU; Drug: Ipatasertib; Drug: Leucovorin; Drug: Oxaliplatin
- Arm B (mFOLFOX + Ipat 600mg) (Experimental): Participants received ipatasertib at a dose of 600mg once daily for 7 consecutive days (beginning on Day 1) in combination with mFOLFOX6 chemotherapy (comprising of oxaliplatin, leucovorin, and 5-FU) on Day 1, in 14-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: 5-FU; Drug: Ipatasertib; Drug: Leucovorin; Drug: Oxaliplatin
- Arm C (Pac + Ipat 400mg) (Experimental): Participants received ipatasertib at a dose of 400mg once daily for 21 consecutive days (beginning on Day 1) in combination with paclitaxel on Days 1, 8, and 15, in 28-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Arm C (Pac + Ipat 600mg) (Experimental): Participants received ipatasertib at a dose of 600mg once daily for 21 consecutive days (beginning on Day 1) in combination with paclitaxel on Days 1, 8, and 15, in 28-day continuous cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Arm D (Enza + Ipat 400mg) (Experimental): Participants received ipatasertib at a dose of 400mg once daily alone for 8 days, then from Day 9, ipatasertib will be administered in combination with enzalutamide once daily for 27 days (Cycle 1 duration = 35 days). Participants received both ipatasertib and enzalutamide once daily continuously in subsequent 28-days cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first. Higher (up to 600 mg) or lower dose of ipatasertib may be evaluated in subsequent cycles depending upon safety, tolerability, and pharmacokinetics of the first cycle.
  Interventions: Drug: Enzalutamide; Drug: Ipatasertib
- Arm D (Enza + Ipat 600mg) (Experimental): Participants received ipatasertib at a dose of 600mg once daily alone for 8 days, then from Day 9, ipatasertib will be administered in combination with enzalutamide once daily for 27 days (Cycle 1 duration = 35 days). Participants received both ipatasertib and enzalutamide once daily continuously in subsequent 28-days cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first. Higher (up to 600 mg) or lower dose of ipatasertib may be evaluated in subsequent cycles depending upon safety, tolerability, and pharmacokinetics of the first cycle.
  Interventions: Drug: Enzalutamide; Drug: Ipatasertib
- Arm D (Enza + Ipat 400-600mg) (Experimental): Participants received ipatasertib at a dose of 400-600mg once daily alone for 8 days, then from Day 9, ipatasertib will be administered in combination with enzalutamide once daily for 27 days (Cycle 1 duration = 35 days). Participants received both ipatasertib and enzalutamide once daily continuously in subsequent 28-days cycles, until disease progression, unacceptable toxicity, or use of another anti-cancer therapy, whichever occurred first. Higher (up to 600 mg) or lower dose of ipatasertib may be evaluated in subsequent cycles depending upon safety, tolerability, and pharmacokinetics of the first cycle.
  Interventions: Drug: Enzalutamide; Drug: Ipatasertib

INTERVENTIONS:
Drug: 5-FU — 5-FU at a dose level of 400 mg/m^2 as intravenous (IV) injection followed by a dose of 2400 mg/m^2 as IV infusion over 46 hrs will be administered on Day 1 of each 14-day cycle until disease progression or unacceptable toxicity.
  Other Names: Adrucil
  Arms: Arm B (mFOLFOX + Ipat 100mg); Arm B (mFOLFOX + Ipat 200mg); Arm B (mFOLFOX + Ipat 400mg); Arm B (mFOLFOX + Ipat 600mg)
Drug: Docetaxel — Docetaxel will be administered at dose level of 75 mg/m^2 as IV infusion over 1 hr on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Arms: Arm A (Doc + Ipat 100mg); Arm A (Doc + Ipat 200mg); Arm A (Doc + Ipat 400mg); Arm A (Doc + Ipat 600mg)
Drug: Enzalutamide — Enzalutamide will be administered orally at a dose level of 160 mg once daily continuously as per schedule defined in respective arm until disease progression or unacceptable toxicity.
  Arms: Arm D (Enza + Ipat 400-600mg); Arm D (Enza + Ipat 400mg); Arm D (Enza + Ipat 600mg)
Drug: Ipatasertib — Ipatasertib will be administered orally (in escalating doses during Stage 1 followed by at a dose decided during Stage 1) as per schedule defined in the respective arms.
Drug: Leucovorin — Leucovorin at a dose level of 400 mg/m^2 as IV infusion over 2 hrs will be administered on Day 1 of each 14-day cycle until disease progression or unacceptable toxicity.
  Other Names: Wellcovorin
  Arms: Arm B (mFOLFOX + Ipat 100mg); Arm B (mFOLFOX + Ipat 200mg); Arm B (mFOLFOX + Ipat 400mg); Arm B (mFOLFOX + Ipat 600mg)
Drug: Oxaliplatin — Oxaliplatin at a dose level of 85 mg/m^2 as IV infusion over 2 hours will be administered on Day 1 of each 14-day cycle until disease progression or unacceptable toxicity.
  Other Names: Eloxatin
  Arms: Arm B (mFOLFOX + Ipat 100mg); Arm B (mFOLFOX + Ipat 200mg); Arm B (mFOLFOX + Ipat 400mg); Arm B (mFOLFOX + Ipat 600mg)
Drug: Paclitaxel — Paclitaxel at a dose of 90 mg/m^2 as IV infusion over 1 hr will be administered on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
  Other Names: Taxol
  Arms: Arm C (Pac + Ipat 400mg); Arm C (Pac + Ipat 600mg)

SUMMARY:
This is an open-label, multicenter, Phase Ib, dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics of oral ipatasertib (GDC-0068) administered in combination with either docetaxel (Arm A), or oxaliplatin, leucovorin, 5-fluorouracil (5-FU) (mFOLFOX6 chemotherapy) (Arm B), or paclitaxel (Arm C), in participants with advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective or intolerable. Arm D will assess the safety, tolerability, and pharmacokinetics of ipatasertib administered in combination with enzalutamide in participants with metastatic castration-resistant prostate cancer (CRPC). There will be two stages within each arm of this study: a dose-escalation stage (Stage 1) and a cohort-expansion stage (Stage 2). In Stage 1, approximately 3 to 6 cohorts in Arms A and B and 1 to 2 cohorts in Arms C and D will be evaluated to determine the maximum tolerated dose (MTD) of ipatasertib in a given combination. Additional participants will be enrolled in Stage 2 (cohort expansion), to further characterize the safety and tolerability of ipatasertib in these combinations and to confirm a potential recommended Phase II dose of ipatasertib for each regimen.

NOTE: Arms A, B, and C are closed.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening
* Histologically or cytologically documented advanced or metastatic solid tumors for which established therapy either does not exist or has proven ineffective or intolerable
* Life expectancy greater than or equal to (>=) 12 weeks
* Adequate hematologic and end organ function
* For female participants of childbearing potential and male participants with partners of childbearing potential, agreement (by participant and/or partner) to use highly effective forms of contraception and to continue its use for the duration of the study and for 4 months after last dose of study treatment (for females) and 6 months after last dose of study treatment (for males)

Exclusion Criteria:

* Prior anti-cancer therapy that fulfills the following criteria: a total of more than three (Arms A and B) or two (Arms C and D) prior cytotoxic chemotherapy regimens, high-dose chemotherapy requiring stem-cell support, and irradiation to >=25 percent (%) of bone marrow-bearing areas
* Treatment with chemotherapy, hormonal therapy (except hormone replacement therapy, oral contraceptives, or gonadotropin-releasing hormone (GnRH) agonists or antagonists for prostate cancer), immunotherapy, biologic therapy, radiation therapy (except palliative radiation to bony metastases), or herbal therapy as cancer therapy within 4 weeks prior to initiation of ipatasertib. Exceptions are kinase inhibitors approved by local regulatory authorities, which may be used within 2 weeks prior to initiation of ipatasertib, provided that any clinically-relevant drug-related toxicity has completely resolved and prior approval is obtained from the Medical Monitor
* Palliative radiation to bony metastases within 2 weeks prior to initiation of ipatasertib
* History of Type 1 or Type 2 diabetes requiring regular medication
* Grade >= 2 heart failure or history of unstable angina
* History of clinically significant ventricular arrhythmias or active ventricular arrhythmia requiring medication
* For Arm D only: History of seizure, unexplained loss of consciousness, transient ischemic attack within 12 months of enrollment, cerebral vascular accident, and any brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Arm A: Days 2-21 of Cycle 1 (cycle length=21 days); Arm B: Days 1-14 of Cycles 1 and 2 (cycle length=14 days); Arm C: Days 1-28 of Cycle 1 (cycle length=28 days); Arm D: Days 1-35 of Cycle 1 (cycle length=28 days except for Cycle 1=35 days)
Maximum Tolerated Dose (MTD) of Ipatasertib | Arm A: Days 2-21 of Cycle 1 (cycle length=21 days); Arm B: Days 1-14 of Cycles 1 and 2 (cycle length=14 days); Arm C: Days 1-28 of Cycle 1 (cycle length=28 days); Arm D: Days 1-35 of Cycle 1 (cycle length=28 days except for Cycle 1=35 days)
Recommended Phase II Dose (RP2D) of Ipatasertib | Arm A: Days 2-21 of Cycle 1 (cycle length=21 days); Arm B: Days 1-14 of Cycles 1 and 2 (cycle length=14 days); Arm C: Days 1-28 of Cycle 1 (cycle length=28 days); Arm D: Days 1-35 of Cycle 1 (cycle length=28 days except for Cycle 1=35 days)
Number of Participants With Adverse Events (AEs) | Baseline up until 30 days following the last administration of study treatment or until initiation of another anti-cancer therapy, whichever occurs first (up to a maximum of 9.25 years).

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Docetaxel (Arm A) | Immediately prior to docetaxel infusion, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours (hrs) after start of docetaxel infusion on Day 1 Cycles 1 and 2 (1 cycle=21 days)
Plasma Terminal Half-Life (t1/2) of Docetaxel (Arm A) | Immediately prior to docetaxel infusion, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours (hrs) after start of docetaxel infusion on Day 1 Cycles 1 and 2 (1 cycle=21 days)
Plasma Clearance (CL) of Docetaxel (Arm A) | Immediately prior to docetaxel infusion, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours (hrs) after start of docetaxel infusion on Day 1 Cycles 1 and 2 (1 cycle=21 days)
Volume of Distribution (Vz) of Docetaxel (Arm A) | Immediately prior to docetaxel infusion, 0.5, 1, 1.5, 2, 3, 4, 6, 24 hours (hrs) after start of docetaxel infusion on Day 1 Cycles 1 and 2 (1 cycle=21 days)
Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Total Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Plasma Terminal Half-Life (t1/2) of Total Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Plasma CL of Total Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Vz of Total Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Maximum Observed Plasma Concentration (Cmax) of Total Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Free Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Plasma Terminal Half-Life (t1/2) of Free Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Plasma CL of Free Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Vz of Free Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Maximum Observed Plasma Concentration (Cmax) of Free Platinum (Arm B) | 1, 2, 2.25, 2.5, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Cmax of 5-FU (Arm B) | 2, 2.25, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Steady-State Concentration (Css) of 5-FU (Arm B) | 2, 2.25, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) of 5-FU (Arm B) | 2, 2.25, 3, 4, 6, 24, 48 hrs after ipatasertib Day 1 dose in Cycle 1 (1 cycle=14 days)
Cmax of Paclitaxel (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
Cmax of Paclitaxel Metabolite (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
AUC(0-inf) of Paclitaxel (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
AUC(0-inf) of Paclitaxel Metabolite (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
Plasma CL of Paclitaxel (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
Plasma CL of Paclitaxel Metabolite (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
Vz of Paclitaxel (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
Vz of Paclitaxel Metabolite (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
Plasma t1/2 of Paclitaxel (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
Plasma t1/2 of Paclitaxel Metabolite (Arm C) | 1, 2, 3, 4, 6, 24 hrs after ipatasertib Day 8 dose in Cycle 1 (1 cycle=28 days)
AUC(0-24) of Enzalutamide (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
AUC(0-24) of Enzalutamide Metabolite (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Time to Reach Cmax (Tmax) of Enzalutamide (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Tmax of Enzalutamide Metabolite (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Cmax at Steady State (Cmax,ss) of Enzalutamide (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Cmax,ss of Enzalutamide Metabolite (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
AUC(0-24) of Ipatasertib (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
AUC(0-24) of Ipatasertib Metabolite (G037720) (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Tmax of Ipatasertib (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Tmax of Ipatasertib Metabolite (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Cmax,ss of Ipatasertib (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Cmax,ss of Ipatasertib Metabolite (Arm D) | Day 8 Cycle 1,2 and Day 1 Cycle 3: Immediately prior to ipatasertib dose, 1,2,3,4,6,24 hours post dose (Cycle=28 days except for Cycle 1=35 days)
Tmax of Ipatasertib (Arm A) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS on Day 2 Cycle 1 (1 cycle=21 days)
Tmax of Ipatasertib (Arm B) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS Day 1 Cycle 1 (1 cycle=14 days)
Tmax of Ipatasertib (Arm C) | PRDS, 1, 2, 3, 4, 6, 24 hrs PSDS Day 8 Cycle 1 (1 cycle=28 days)
Tmax of Ipatasertib Metabolite (Arm A) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS on Day 2 Cycle 1 (1 cycle=21 days)
Tmax of Ipatasertib Metabolite (Arm B) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS Day 1 Cycle 1 (1 cycle=14 days)
Tmax of Ipatasertib Metabolite (Arm C) | PRDS, 1, 2, 3, 4, 6, 24 hrs PSDS Day 8 Cycle 1 (cycles=21 days, Cycle 1=35 days)
Cmax,ss of Ipatasertib (Arm A) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS on Day 2 Cycle 1 (1 cycle=21 days)
Cmax,ss of Ipatasertib (Arm B) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS Day 1 Cycle 1 (1 cycle=14 days)
Cmax,ss of Ipatasertib (Arm C) | PRDS, 1, 2, 3, 4, 6, 24 hrs PSDS Day 8 Cycle 1 (1 cycle=28 days)
Cmax,ss of Ipatasertib Metabolite (Arm A) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS on Day 2 Cycle 1 (1 cycle=21 days)
Cmax,ss of Ipatasertib Metabolite (Arm B) | PRDS, 0.5, 1, 2, 3, 4, 6, 24 hrs PSDS Day 1 Cycle 1 (1 cycle=14 days)
Cmax,ss of Ipatasertib Metabolite (Arm C) | PRDS, 1, 2, 3, 4, 6, 24 hrs PSDS Day 8 Cycle 1 (1 cycle=28 days)
Number of Participants With Objective Response as Determined by Investigator Review of Tumor Assessments Using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Baseline up to disease progression or death, whichever occurs first (up to approximately 6 years)
Duration of Response (DOR) as Determined by Investigator Review of Tumor Assessments Using RECIST v1.1 | Baseline up to disease progression or death, whichever occurs first (up to approximately 6 years)
Progression-free Survival (PFS) as Determined by Investigator Review of Tumor Assessments Using RECIST v1.1 | Baseline up to disease progression or death, whichever occurs first (up to approximately 6 years)
Radiographic Progression-free Survival (rPFS) as Determined by Investigator (Arm D only) | Baseline up to radiographic disease progression or death, whichever occurs first (up to approximately 6 years)
Time to Treatment Failure (TTF) | Baseline up to treatment discontinuation for any reason (up to approximately 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Maslyar, M.D., Study Director — Genentech, Inc.
Locations (11):
- United States (7):
  - California Pacific Med Center, San Francisco, California
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - SCRI, Nashville, Tennessee
  - Virginia Oncology Associates, Norfolk, Virginia
- Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif, France
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico Universitario de Valencia, Valencia
- The Royal Marsden Hospital, Sutton, United Kingdom

REFERENCES:
- [Derived] Isakoff SJ, Tabernero J, Molife LR, Soria JC, Cervantes A, Vogelzang NJ, Patel MR, Hussain M, Baron A, Argiles G, Conkling PR, Sampath D, Maslyar D, Patel P, Chan W, Gendreau S, Musib L, Xu N, Ma H, Lin K, Bendell J. Antitumor activity of ipatasertib combined with chemotherapy: results from a phase Ib study in solid tumors. Ann Oncol. 2020 May;31(5):626-633. doi: 10.1016/j.annonc.2020.02.007. Epub 2020 Feb 20. PMID 32205017